CLINICAL TRIAL: NCT06622122
Title: Exploring the Mechanism of Mindfulness Intervention: Manipulating the Dose of Cognitive Flexibility Intervention
Brief Title: Mechanisms of Mindfulness Intervention: Cognitive Flexibility Dose Manipulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xinghua Liu, Director, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E20240925
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Emotional Distress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- MIED group (Experimental): Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge, and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression, and other emotional problems.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version
- MIED+CF group (Experimental): The increase in cognitive flexibility dosage involves incorporating additional psychoeducational content related to cognitive flexibility and corresponding exercises to enhance cognitive flexibility within the MIED (Mindfulness Intervention for Emotional Distress) program.
  Interventions: Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-increase cognitive flexibility
- waitlist control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-normal version — Mindfulness Intervention for Emotional Distress (MIED) program provides standard audio instructions for mindfulness exercises, introduces the nature and law of anxiety, depression, and other emotions, the source of anxiety, depression, and other emotional distress, and the strategies and methods to alleviate emotional distress. These exercises, knowledge and strategies are based on the latest progress in the field of psychological counseling and treatment, and their application in daily life can help alleviate anxiety, depression and other emotional problems.
  Arms: MIED group
Behavioral: Mindfulness Intervention for Emotional Distress(MIED)-increase cognitive flexibility — Increase the intervention dose of cognitive flexibility in Mindfulness Intervention for Emotional Distress (MIED). For example, including more cognitive reappraisal practice, psychoeducational content and practice about regarding thoughts just as thoughts.
  Arms: MIED+CF group

SUMMARY:
This study hopes to:

1. explore whether an increase in the dosage of cognitive flexibility intervention corresponds to greater effectiveness of mindfulness intervention in alleviating emotional distress.
2. explore whether cognitive flexibility mediates the effects of mindfulness intervention on alleviating emotional distress.

DETAILED DESCRIPTION:
Epidemiological findings in "The Lancet Psychiatry" indicated that anxiety disorders, including generalized anxiety disorder, panic disorder, and social anxiety disorder, are the most prevalent category of disorders in China, with a lifetime prevalence of 7.6%. Depression follows closely with a lifetime prevalence of 6.8%. With the outbreak of the COVID-19 pandemic in 2020, the prevalence of both anxiety and depressive disorders increased. However, the current availability of psychological intervention resources in China is inadequate to meet the demand. This underscores the critical importance of developing effective and efficient psychological intervention approaches, as well as investigating their effectiveness and mechanisms to optimize intervention strategies.

Epidemiological findings in "The Lancet Psychiatry" indicated that anxiety disorders, including generalized anxiety disorder, panic disorder, and social anxiety disorder, are the most prevalent category of disorders in China, with a lifetime prevalence of 7.6%. Depression follows closely with a lifetime prevalence of 6.8%. With the outbreak of the COVID-19 pandemic in 2020, the prevalence of both anxiety and depressive disorders increased. However, the current availability of psychological intervention resources in China is inadequate to meet the demand. This underscores the critical importance of developing effective and efficient psychological intervention approaches, as well as investigating their effectiveness and mechanisms to optimize intervention strategies.

In recent years, mindfulness-based interventions (MBIs) have been increasingly applied to alleviate emotional distress in both clinical and non-clinical populations, with their efficacy widely supported. Additionally, numerous researchers have explored the mechanisms underlying mindfulness and MBIs, proposing various theories. One of the mechanisms frequently suggested by researchers is cognitive flexibility. However, there has been limited direct investigation into the mechanisms of cognitive flexibility and its related processes or abilities. Cognitive flexibility (CF) is considered a common etiological factor or transdiagnostic characteristic of emotional distress, including anxiety and depression. Nevertheless, few studies have explored the mechanisms of how mindfulness interventions alleviate emotional distress from the perspective of cognitive flexibility and the transdiagnostic characteristics of anxiety and depression. This lack of research hampers our ability to obtain sufficient information to develop or enhance mindfulness-based intervention methods to assist individuals with emotional disorders or highly emotionally distressed subclinical populations.

This study is grounded in the critical role of CF in the generation and maintenance of emotional distress, as well as the mindfulness principle of approaching pain with awareness and acceptance (non-judgmental and non-reactive). It posits that cognitive flexibility might be a potential mechanism through which mindfulness interventions alleviate emotional distress. Following the criteria for establishing mechanisms, this research investigates this issue. Based on the current state of research, cognitive flexibility as a mechanism for MBIs to alleviate emotional distress meets the plausibility criterion and partially satisfies the strong association criterion and experimental manipulation criterion. However, further research is needed to assess its consistency criterion, temporal precedence criterion, and gradient criterion.

The current study primarily focuses on the experimental manipulation and gradient criteria. The aim is to examine whether the mechanism of cognitive flexibility meets the experimental manipulation and gradient criteria by adjusting the content of the mindfulness intervention for emotional distress (MIED) program, which can directly impact distress tolerance and manipulate the dosage of cognitive flexibility intervention.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects with scores greater than 21 on the Kessler Psychological Distress Scale.
* - Aged 18-65 years old.

Exclusion Criteria:

* - Subjects who could not access the Internet;
* - Subjects with insufficient Chinese ability;
* - Subjects who have participated in mindfulness based projects for more than 6 weeks before, and / or the current frequency of meditation practice is more than once a week;
* - Subjects with schizophrenia or psychotic affective disorder, current organic mental disorder, substance abuse disorder and generalized developmental disorder;
* - Subjects with high risk of suicide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-11 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-11 (Estimated)

PRIMARY OUTCOMES:
Weekly changes of Five Facet Mindfulness Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  The Five Facet Mindfulness Questionnaire is a self-reported questionnaire measuring mindfulness levels. Scores range from 39 to 195, with higher scores indicating higher levels of mindfulness.
Weekly changes of 10-item Kessler Psychological Distress Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  The 10-item Kessler Psychological Distress Scale is a self-reported questionnaire measuring distress. Scores range from 10 to 50, with higher scores indicating higher levels of distress.
Weekly changes of Rumination-Reflection Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  Rumination-Reflection Questionnaire is a self-reported questionnaire measuring Rumination level.Scores range from 12 to 60, with higher scores indicating higher levels of Rumination.
Weekly changes of Emotion Regulation Questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  Emotion Regulation Questionnaire is a self-reported questionnaire measuring cognitive reappraisal level.Scores range from 6 to 42, with higher scores indicating higher levels of cognitive reappraisal ability.
Weekly changes of Overall Anxiety Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  The Overall Anxiety Severity and Impairment Scale is a self-reported questionnaire measuring anxiety. Scores range from 0 to 20, with higher scores indicating higher levels of anxiety.
Weekly changes of Overall Depression Severity and Impairment Scale during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  The Overall Depression Severity and Impairment Scale is a self-reported questionnaire measuring depression. Scores range from 0 to 20, with higher scores indicating higher levels of depression.
Weekly changes of Cognitive flexibility Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  Cognitive flexibility Inventory is a self-reported questionnaire measuring Cognitive flexibility level.Scores range from 20 to 100, with higher scores indicating higher levels of Cognitive flexibility.
Weekly changes of experiences questionnaire during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  experiences questionnaire is a self-reported questionnaire measuring decentralization ability. Scores range from 20 to 100, with higher scores indicating higher levels of Decentralized ability.
Weekly changes of Beck Anxiety Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  Beck Anxiety Inventory is a self-reported questionnaire measuring Anxiety level.Scores range from 0 to 63, with higher scores indicating higher levels of Anxiety.
Weekly changes of Beck Depression Inventory during the intervention | pre-intervention; weekly during the 7-week intervention; immediately after the intervention
  Beck Depression Inventory is a self-reported questionnaire measuring depression level.Scores range from 0 to 63, with higher scores indicating higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xinghua Liu, Principal Investigator — School of Psychological and Cognitive Sciences, Peking University
Locations (1):
- Peking University, Beijing, China

IPD SHARING:
Plan to Share IPD: No